CLINICAL TRIAL: NCT00499902
Title: Phase 2, Multicenter, Open-Label, Two-Stage Study to Evaluate the Safety and Efficacy of Intra-Arterial Catheter-Directed Alfimeprase for Restoration of Neurologic Function and Rapid Opening of Arteries in Stroke (CARNEROS-1)
Brief Title: Phase 2 Proof-of-Concept Study of the Safety and Efficacy of Alfimeprase to Rapidly Open Arteries and Restore Brain Function Following a Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: CO Phase 2 data did not show sufficient improvement in cath opening at higher dose/concentration evaluated. Nuvelo ended further clinical dev of alfimeprase.
Sponsor: ARCA Biopharma, Inc. (Industry)
Responsible Party: Brian Kersten, PhD, Nuvelo, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HA009
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Acute Ischemic Stroke
Keywords: AIS; acute ischemic stroke; stroke; alfimeprase; blood clot; brain; thrombus; thrombolytic; thrombosis; plasminogen activator; arterial flow; neurology; intra-arterial; intra-thrombus; catheter-directed; symptomatic ICH; ICH; AOL; arterial occlusive lesion; recanalization
MeSH Terms: conditions — Ischemic Stroke; Stroke; Thrombosis | interventions — alfimeprase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 stages (Other): This is a two-stage study. The first stage is in a three-tier dose escalation format, followed by a second stage during which subjects will be randomized in an equal proportion to up to 3 qualifying dose arms.
  Interventions: Drug: alfimeprase

INTERVENTIONS:
Drug: alfimeprase — Alfimeprase will be given as a single bolus of 1mg/2mL, or a split bolus of 5mg/2mL or 10mg/2mL in a three-tier dose escalation format. The 5mg and 10mg doses will be administered as split doses with 1/2 of the total dose given initially and 1/2 of the total dose given 30 minutes after the initial dose.

SUMMARY:
The purpose of this study is to identify a safe and effective bolus dose of intra-arterial/intra-thrombus alfimeprase in acute ischemic stroke (AIS) 3 to 9 hours from symptom onset.

DETAILED DESCRIPTION:
Currently approved drug therapy for AIS is limited by the need to treat within 3 hours of symptom onset. Alfimeprase acts to degrade fibrin directly and is inactivated locally by circulating alpha-2 macroglobulin. This study will determine whether treatment with alfimeprase facilitates rapid restoration of arterial blood flow with avoidance of symptomatic hemorrhagic conversion in subjects with AIS within 3 to 9 hours of symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of AIS defined as the sudden onset of an acute focal neurological deficit presumed to be due to cerebral ischemia
* Arterial occlusion of the carotid T or a M1, M2, or M1-M2 branch of the middle cerebral artery (MCA) as documented by CT angiography or magnetic resonance angiography
* Arteriographically confirmed occlusion of the carotid T or a M1, M2, or M1-M2 branch of the MCA
* The subject (or legally acceptable representative) must give written informed consent
* Age 18 years to 85 years
* Onset of symptoms of AIS (i.e., last known well time) within 3-9 hours
* Baseline NIHSS of 4 to 25
* Available for follow-up assessments at 30 and 90 days

Exclusion Criteria:

* Contraindication to systemic anticoagulation including any history of prior intracranial hemorrhage
* Uncontrolled hypertension at study entry as defined by systolic blood pressure greater than 180 mmHg or diastolic blood pressure greater than or equal to 100 mmHg on repeated measures prior to study entry despite the use of IV antihypertensive agents
* Expectation based on timing of presentation that alfimeprase administration will not be able to be completed by 9 hours after stroke onset
* Inability to initiate alfimeprase within 120 minutes of the qualifying imaging scan
* Coma
* Rapidly improving neurological symptoms at the time of screening
* Brain CT or MRI evidence of intracranial bleeding of any age
* High clinical suspicion for subarachnoid hemorrhage despite a negative baseline CT or MRI
* CT evidence of an acute and/or evolving hypodensity greater than 1/3 of the MCA territory in the vascular territory to be treated or Alberta Stroke Program Early CT Score (ASPECTS) of less than or equal to 5
* MRI diffusion weighted imaging lesion greater than 1/3 of the MCA territory in the vascular distribution to be treated
* Carotid artery and/or intracranial artery stenosis that precludes safe passage of a microcatheter to treat the primary AOL
* Life expectancy of less than 6 months
* History of significant acute or chronic kidney disease, including known nephrotic syndrome, that would preclude safe contrast angiography
* Known allergy to contrast agents
* History of immune deficiency
* History of heparin-induced thrombocytopenia
* Participation in any study of an investigational device, medication, biologic, or other agent within 30 days prior to enrollment (Stage I)/randomization (Stage II)
* Any stroke, myocardial infarction, or use of thrombolytic therapy (including investigational thrombolytic therapy) within 3 months prior to enrollment (Stage I)/randomization (Stage II)
* Past participation in any alfimeprase clinical trial
* Pregnant, lactating, or actively menstruating women and women of child-bearing potential who are not using adequate contraceptive precautions
* Current use of oral anticoagulants or an international normalized ratio (INR) greater than 1.4
* Any non-atherosclerotic arteriopathy
* Any prior neurologic event that would obscure the radiographic or clinical evaluation of the new index neurological deficits
* Subjects with known renal insufficiency defined as a serum creatinine >2 mg/dL (>180 mmoL/L)
* Subjects with known clinically significant hepatic disease defined as transaminase values > 3x upper limit of normal
* Subjects with any malignant neoplasm diagnosed within five years prior to screening, with the exception of basal cell carcinoma of the skin and fully resected squamous cell carcinoma of the skin
* Subjects with a platelet count less than 100,000/mm3
* Subjects with a baseline serum glucose level less than 50 mg/dL or greater than 300 mg/dL
* Subjects receiving any dose of a heparinoid or a non-prophylactic intensity dose of a low molecular weight heparin within the 24-hour period prior to study drug administration
* Any other subject feature that in the opinion of the investigator should preclude study participation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-06; Primary Completion 2008-05 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Symptomatic intracerebral hemorrhage (ICH) defined as a greater than or equal to 4-point increase in NIHSS compared to baseline at the time of CT evidence of ICH within 24 hours of study drug administration.
Recanalization of primary arterial occlusive lesion (AOL) using the Thrombolysis in Myocardial Infarction (TIMI) classification; a score of II or III will be considered success.

SECONDARY OUTCOMES:
Relative hypotension requiring treatment (i.e. volume expanders and/or vasopressors)
New cardiac events (e.g., cardiac ischemia, congestive heart failure, and dysrhythmia)
Relative hypotension not requiring treatment
Major bleeding events (TIMI definition)
Hemorrhagic transformation: hemorrhagic infarction (Type 1 and 2), parenchymal hematoma formation (Type 1 and 2)
Intracerebral hemorrhage outside of the stroke territory
New AIS
AEs/SAEs/All cause mortality
Changes in chemistry, hematology, coagulation, and alpha-2-macroglobulin parameters based on central laboratory measurements
Anti-alfimeprase antibody detection based on central laboratory measurements
Recanalization of the primary AOL
Global reperfusion of the primary AOL distal vascular bed defined by the Thrombolysis in Cerebral Infarction (TICI) score
Neurological benefit as assessed by individual and combined analysis of NIHSS, mRS, and BI

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Begelman, MD, Study Director — ARCA Biopharma, Inc.
Locations (21):
- United States (16):
  - UCLA Medical Center, Los Angeles, California
  - Northwestern Medical Center, Chicago, Illinois
  - Ruan Neurology & Clinical Research Center, Des Moines, Iowa
  - University of Iowa Hospital, Iowa City, Iowa
  - University of Kansas School of Medicine, Via Christi Regional Medical Center, Wichita, Kansas
  - Norton Hospital, Louisville, Kentucky
  - Michigan State University, Sparrow Hospital, Lansing, Michigan
  - Albany Medical Center Hospital, Albany, New York
  - Kalieda Health, MFH, Buffalo, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Oregon Stroke Center, Portland, Oregon
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Canada (5):
  - University of Calgary, Foothills Medical Centre, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Trilium Health Center, Mississauga, Ontario
  - University Health Network Toronto, Toronto, Ontario
  - Montreal Neurological Institute, Montreal, Quebec

REFERENCES:
- See also: Company Website — http://www.Nuvelo.com